CLINICAL TRIAL: NCT02893059
Title: Evaluation of a Data Collection Tool in Clinical Research: Comparison Between the Data Collected by Patient Diary and Data From Medical Administrative Databases
Acronym: CORD
Status: Withdrawn | Type: Observational
Why Stopped: the investigator has left the facility
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC/2014/CC-01
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Case Report Form; Declaration Bias; Health Insurance Database

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to estimate the reporting bias of patients in terms of prescripted drug and care consumption by comparing data collected in a patient diary and database of health insurance .

ELIGIBILITY:
Inclusion Criteria:

* incident and prevalent cases of patients with type I or type II diabetes. arthritis:
* incident and prevalent cases of rheumatoid arthritis patients defined according to the ACR-EULAR criteria 2010 (Aletaha D et al, 2010).

Renal failure :

• incident and prevalent cases of patients with kidney disease stage 3 or 4, transplanted or not.

Prostate cancer :

• Incident cases of patients with prostate cancer regardless of the stage at diagnosis (positive prostate biopsy).

Breast cancer :

• Incident cases of patients with breast cancer regardless of the stage at diagnosis (biopsy positive breast).

Colorectal cancer :

• Incident cases of patients with colorectal cancer regardless of the stage at diagnosis (colonoscopy and polyp biopsy positive).

Exclusion Criteria:

- The subject participates in an experimental study of research affecting the therapeutic management of the patient.

* The subject is exclusion period determined by a previous study.
* The subject is under judicial protection, guardianship or curatorship.
* It is not possible to give informed about information
* The subject does not read French and is not autonomous filling a questionnaire.
* The patient has psychiatric disorders.
* The subject is an emergency.
* Monitoring between patient visits than 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of incident and prevalent cases of patients with chronic disease (diabetes, rheumatoid arthritis, chronic renal failure) or incident cases of prostate cancer, breast cance or colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
comparison of data collected in a patient diary and data stored in the database of health insurance | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: christel castelli, PhD, Study Director — CHU Nimes